CLINICAL TRIAL: NCT00566800
Title: Chemoprevention Trial Using Erlotinib in Barrett's Esophagus With High-Grade Dysplasia
Brief Title: Erlotinib in Treating Patients With Barrett Esophagus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000576425; VAMCK-JB0027; GENENTECH-OSI3717s
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2008-01

CONDITIONS: Esophageal Cancer; Precancerous Condition
Keywords: esophageal cancer; Barrett esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Precancerous Conditions; Barrett Esophagus | interventions — Erlotinib Hydrochloride; Biopsy

INTERVENTIONS:
Drug: erlotinib hydrochloride
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. Erlotinib may keep esophageal cancer from forming in patients with Barrett esophagus by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with Barrett esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if erlotinib hydrochloride can be used as a chemopreventive agent that can cause histologic regression of Barrett esophagus in patients at high risk of developing esophageal cancer associated with high-grade dysplasia.

Secondary

* To assess whether erlotinib hydrochloride can cause molecular alterations in EGFR, phospho-EGFR, cyclin D1, cdc2, p16, p53, PCNA, COX-2, and ploidy in Barrett esophagus with high-grade dysplasia.
* To establish surrogate markers of chemoprevention in Barrett esophagus with high-grade dysplasia.
* To validate the histologic scoring of Barrett dysplasia developed by our group.
* To evaluate toxicities associated with the use of erlotinib hydrochloride in patients with Barrett esophagus associated with high-grade dysplasia.

OUTLINE: Patients receive oral erlotinib hydrochloride once daily for 3 months. Patients showing no evidence of progression to cancer by esophagogastroduodenoscopy (EGD) with biopsy receive an additional 3 months of treatment. All patients then undergo repeat EGD, biopsy, and determination of molecular markers (i.e., EGFR, phospho-EGFR, cyclin D1, cdc2, p16, p53, PCNA, COX-2, and ploidy).

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Barrett esophagus with high-grade dysplasia
* Refused surgery or other localized therapy for high-grade dysplasia
* No invasive esophageal carcinoma

PATIENT CHARACTERISTICS:

* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST and ALT < 3 times upper limit of normal (ULN)
* Alkaline phosphatase < 3 times ULN
* No uncontrolled medical condition
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 1 week after completion of study treatment
* Able to swallow tablets or dissolved tablets
* No known hypersensitivity to erlotinib hydrochloride
* No symptoms suggestive of malignancy (e.g., weight loss or vomiting)
* No history of other malignancies
* No uncontrolled medical or psychiatric condition that would preclude treatment under this clinical trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior exposure to erlotinib hydrochloride
* No concurrent antineoplastic or antitumor agents, including chemotherapy, radiotherapy, immunotherapy, or hormonal therapy
* No concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
Histologic regression of Barrett esophagus with high-grade dysplasia by chemoprevention with erlotinib hydrochloride

SECONDARY OUTCOMES:
Molecular alterations in EGFR, phospho-EGFR, cyclin D1, cdc2, p16, p53, PCNA, COX-2, and ploidy
Validation of histologic scoring of Barrett dysplasia
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Joaquina C. Baranda, MD, Principal Investigator — Kansas City Veteran Affairs Medical Center
Locations (1):
- Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri, United States